CLINICAL TRIAL: NCT03325725
Title: Intra-laryngeal Implant for Treatment of Chronic Aspirations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Competent Authority did not give the authorization to start the study.
Sponsor: ProTiP Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NB_LD
Record Dates: First submitted 2017-10-17; First posted 2017-10-30 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Aspiration Pneumonia; Tracheostomy Complication
Keywords: severe aspiration
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NewBreez LD Intra-laryngeal implant (Experimental)
  Interventions: Device: NewBreez LD intra-laryngeal implant

INTERVENTIONS:
Device: NewBreez LD intra-laryngeal implant — NewBreez LD intra-laryngeal implantation

SUMMARY:
This study evaluates the medical device Newbreez LD is designed to protect the lower airways from saliva, liquids and food aspirations in tracheotomized patients suffering from chronic aspirations that require specific care and may lead to complications, including inhalation pneumonia.

DETAILED DESCRIPTION:
Patients suffering from swallowing disorders characterized by chronic aspirations (repeated episodes of aspirations defined as penetration of material - liquids, food, saliva, into the respiratory system due to a malfunctioning of the swallowing mechanism) are subject to pathologies and pulmonary insufficiencies. The risks of aspiration pneumonia or suffocation are significantly greater if the patient is not able to expectorate and thus engages the vital prognosis. There are several methods to treat chronic aspirations: the least invasive methods involve adopting postures and/or positions of the body during swallowing and adapting food textures; when these treatments are insufficient there is the need to recur to more advanced ones to protect the airways and keep the patient on a sufficient nutrition.

For these severe cases, heavier surgical methods can be also considered. These methods lead to important anatomical changes, with a variable degree of reversibility, up to irreversibility (eg total laryngectomy). Among surgical methods, there is also an implant of a tracheotomy cuffed cannula that allows patient to breathe through a hole in the trachea. The efficacy of this solution is highly controversial as reported by numerous studies and several adverse effects are reported on the tracheal duct.

Due to the interest of a prosthetic treatment and the disadvantages of the current methods and devices, PROTiP Medical has developed a closed intra-laryngeal implant: NewBreez LD. This device is innovative because its geometry has been optimized to conform totally to the anatomy of the larynx with the aim to ensure a sealing against saliva, liquids and food aspirations.

ELIGIBILITY:
Inclusion Criteria:

* Swallowing disorders characterized by chronic aspirations;
* Tracheotomy performed, inter alia, in the management of swallowing disorders;
* Aged over 18;
* Willing and able to comply with the requirements of the study;
* Informed consent signed;
* Affiliated patient or beneficiary of the social security system.

Exclusion Criteria:

* Do not implant in patients with incomplete cricoid cartilage (surgery or other);
* Do not implant in patients with tracheotomy performed by cricothyroidectomy or between cricoid cartilage and the 1st tracheal ring;
* Do not implant in patients with tracheal lumen in the 1st tracheal ring, the lateral and anteroposterior diameters of which are less than 11 mm;
* Do not implant in patients with tight trismus;
* Do not implant in subjects less than 18 years of age;
* Do not implant in patients with bleeding disorders;
* Do not implant in patients contraindicated to general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Sealing of the NewBreez LD: Protection of the lower airways will be assessed using the gold standard exam, videofluoroscopy (VFS) | 7 days
  Protection of the lower airways will be assessed using the gold standard exam, videofluoroscopy (VFS)

OTHER OUTCOMES:
Stability of the NewBreez LD: Number of patients who kept the implant until the end of the study period. | 30 days
  Number of patients who kept the implant until the end of the study period.
Safety of the NewBreez LD: Number of patient with adverse events will be assessed at each follow-up during the study period | 2, 7, 30 days
  Number of patient with adverse events will be assessed at each follow-up during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Christian Debry, Pr., Principal Investigator — CHU Strasbourg
Locations (2):
- France (2):
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse